CLINICAL TRIAL: NCT07034092
Title: Feasibility Study to Evaluate the Safety and Efficacy of the ePATH System for endoAVF Creation
Brief Title: PATH-03 Paraguay Feasibility Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pathfinder Medical (Industry)
Collaborators: MINSA SA (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SKL-TF60000 10.4; Pathfinder Medical (Other: The study is funded only by Pathfinder Medical and is not listed in any other databases.)
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Kidney Disease, End-Stage
Keywords: fistula, AVF, endoAVF, hemodialysis, vascular access; endovascular AVF
MeSH Terms: conditions — Kidney Failure, Chronic; Fistula

STUDY DESIGN:
Intervention Model Description: An endoAVF for dialysis access will be created in the treated subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): An endoAVF will be created in the treated subjects.
  Interventions: Device: ePATH System will be used to create an endoAVF

INTERVENTIONS:
Device: ePATH System will be used to create an endoAVF — An endoAVF will be created in subjects that need fistulas for hemodialysis

SUMMARY:
The goal of this study is to evaluate the safety and effectiveness of the ePATH system in the creation of an endovascular AVF (endoAVF) in patients who require or will soon require hemodialysis and are eligible for a fistula.

ELIGIBILITY:
Inclusion Criteria:

1. Patients deemed eligible for creation of an AV fistula according to institutional or local guidelines and/or clinical judgement of the investigator
2. Adults (age >18 years old)
3. Non-reversible kidney failure requiring hemodialysis (this can include pre-dialysis patients)
4. Target vein diameter of ≥2.0 mm
5. Target artery diameter of ≥2.0 mm
6. Both radial and ulnar artery flow to the hand, confirmed with Duplex Ultrasound and/or Allen's test (i.e. palmar arch)
7. Able to provide informed consent
8. Able to comply with follow-up visit assessment requirements
9. Patient is free from clinically significant conditions or illnesses that might compromise the procedure or the AVF

Exclusion Criteria:

1. Significant central venous stenosis or narrowing that exceeds 50% based on imaging
2. Hypercoagulable state or known bleeding diathesis
3. NHYA Class III or IV heart failure
4. Estimated life-expectancy of <1 year based on the physician's opinion
5. Oedema of extremities
6. Current diagnosis of carcinoma
7. Pregnant or breastfeeding women
8. Diagnosed or suspected skin disease at the access site
9. Immunosuppression or otherwise immunocompromised patients
10. Currently being treated with another investigational device or medication
11. Allergy to contrast or other drugs associated with surgery, e.g., sedation agents, or to device materials
12. Anatomy that prevents formation of AVF, e.g., misalignment of vessels or tortuosity
13. Patient is unwilling to undergo 2nd stage procedure, e.g. endovascular prothesis placement or balloon dilatation, if required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 3 months
  Proportion of patients that experience one or more serious ePATH device-related or ePATH portion of the procedure-related adverse events during the first 3 months following AVF creation.

SECONDARY OUTCOMES:
Technical Success | 7 days
  Technical success: Successful creation of a fistula with the ePATH system. Verification that an endoAVF has been created with the ePATH system and that it remains patent 1-7 days after the index procedure. Patency will be defined by an experienced examiner as the presence of a bruit as detected by stethoscope, or the presence of a thrill, or with duplex ultrasonography for all study endpoints.
AVF maturation | 3 months
  Defined as an AVF that is free from stenosis or thrombosis with an arterial inflow of at least 500 ml/min and/or a diameter of at least 4 mm (as measured by duplex ultrasonography) or the patient was successfully dialysed with 2 needles.
Time to fistula maturation | 3 months
  Number of days between the index procedure and the date at which AVF maturation is achieved
Rate of other device or other procedure-related adverse events | 3 months
  Rate of serious other device (not ePATH device) or other procedure-related (not ePATH portion of the procedure) adverse events at 3 months following the index procedure
Rate of device and/or procedure related infections | 3 months
  Rate of device and/or procedure related infections at 3 months following the index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Adrian A Ebner, MD, Principal Investigator — Sanatorio Italiano
Locations (1):
- Sanatorio Italiano, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No